CLINICAL TRIAL: NCT00561249
Title: Randomized Prospective Trial on the Use of Laser Assisted Hatching (LAH) for Transfer of Frozen/Thawed Embryos in Human IVF/ICSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007/453
Record Dates: First submitted 2007-11-16; First posted 2007-11-20 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: IVF; ICSI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Embryos for transfer are subjected to laser assisted hatching(LAH) following the standard procedure.The LAH procedure lasts two minutes per embryo.
  Interventions: Procedure: laser assisted hatching
- 2 (No Intervention): No intervention

INTERVENTIONS:
Procedure: laser assisted hatching — Embryos for transfer are subjected to laser assisted hatching(LAH) following the standard procedure.The LAH procedure lasts two minutes per embryo
  Arms: 1

SUMMARY:
At the time of transfer of frozen/thawed embryos in human IVF/ICSI, patients are randomized between study and control group.In the control group no additional intervention takes place on the embryos to be transferred,in the study group, embryos for transfer are subjected to laser assisted hatching(LAH) following the standard procedure.The LAH procedure lasts two minutes per embryo.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above
* Female

Exclusion Criteria:

* No exclusion criteria, except not possible to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2007-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
clinical implantation per transferred embryo | fourteen days after transfer

SECONDARY OUTCOMES:
clinical pregnancy and birth per transfer | resp. 12 weeks and 38 weeks after transfer

CONTACTS AND LOCATIONS:
Overall Officials: Petra De Sutter, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be